CLINICAL TRIAL: NCT01532622
Title: Impact of Blueberries on Uric Acid and Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Collaborators: U.S. Highbush Blueberry Council (Other)
Responsible Party: Principal Investigator, Daniel Riche, Associate Professor, University of Mississippi Medical Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2011-0218
Record Dates: First submitted 2012-01-30; First posted 2012-02-14 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: Hyperuricemia
Keywords: Blueberry
MeSH Terms: conditions — Hyperuricemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Blueberry Powder (Active Comparator): Patients will take 30 grams of blueberry powder daily for up to 30 days.
  Interventions: Dietary Supplement: Blueberry Powder
- Placebo Powder (Placebo Comparator): Patients will take 30 grams of placebo powder daily for up to 30 days.
  Interventions: Other: Placebo Powder

INTERVENTIONS:
Dietary Supplement: Blueberry Powder — Patients will take 30 grams of blueberry powder daily for up to 30 days
  Other Names: Blueberry powder from the U.S. Highbush Blueberry Council.
  Arms: Blueberry Powder
Other: Placebo Powder — Patients will take 30 grams of placebo powder daily for up to 30 days.
  Arms: Placebo Powder

SUMMARY:
The purpose of this study is to determine the impact of blueberries on uric acid in patients with hyperuricemia that are not receiving uric acid pharmacotherapy. The central hypothesis the investigators propose is that daily blueberries added to a pre-existing diet will promote uric acid lowering and improve quality of life without detriment to vital signs.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Uric acid > 6.0 mg/dL

Exclusion Criteria:

* Current moderate-to-severe symptomatic gout
* Currently receiving gout pharmacotherapy
* Current participation in another clinical trial
* Documented non-compliance or consistent missed appointments
* Women who are pregnant or nursing

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2012-01; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Change from Baseline and Placebo in Uric Acid Level in Patients Randomized to Treatment Group | Baseline, ~30 days later
  Percent change in uric acid level from baseline after 30 days of treatment with blueberry powder. Since this is designed as a crossover trial, baseline could represent uric acid level at the beginning of the study or after at least a 2-week washout period following placebo administration.

SECONDARY OUTCOMES:
Blood Pressure | Baseline, ~30 days, ~45 days, ~75 days
  Percent change and absolute change of blood pressure from baseline and placebo
Body Weight | Baseline, ~30 days, ~45 days, ~75 days
  Percent change and absolute change of body weight from baseline and placebo
Quality of Life | Baseline, ~30 days, ~45 days, ~75 days
  Quality of life will be assessed using the Health Assessment Questionnaire-Disability Index (HAQ-DI)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Riche, Pharm.D., Principal Investigator — University of Mississippi Medical Center; Marion Wofford, M.D., M.P.H., Principal Investigator — University of Mississippi Medical Center
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States